CLINICAL TRIAL: NCT07313904
Title: Effects of Environmental Fungal Exposure on Bronchial Asthma, Allergic Bronchopulmonary Aspergillosis (ABPA), and Bronchiectasis
Brief Title: Effects of Environmental Fungal Exposure on Bronchial Asthma, ABPA and Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Ningbo University (Network)
Responsible Party: Sponsor
Other Study IDs: 2025-155A-01
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-07

CONDITIONS: Environmental Exposure; Asthma; Bronchiectasis; ABPA
MeSH Terms: conditions — Asthma; Bronchiectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Asthma
- ABPA
- Bronchiectasis
- Healthy control group

SUMMARY:
This study is a prospective, observational study of patients aged 18-80 years with clinical diagnosis of bronchial asthma, allergic bronchopulmonary aspergillosis (ABPA), bronchiectasis and healthy subjects. Among them, the bronchial asthma group will be divided into asthma control group, asthma partial control group and asthma uncontrolled group according to the GINA asthma control classification. Record the baseline information of the subjects in detail, including basic information, disease course, smoking, previous acute attacks and hospitalizations, long-term medication, etc. (including the frequency, dose and duration of ICS use, antifungal drug type, dose, duration of use, and course of treatment), and evaluate and record environmental factors (such as indoor).Humidity, temperature, ventilation, pet keeping, plant planting, etc.) and other lifestyle factors that may affect disease control and fungal exposure. The patient's disease status was assessed using questionnaire scores.

Sputum samples were taken at the time of enrollment.Set (asthma ABPA group uses sputum induction), pulmonary function test and bronchodilator test, FeNO measurement (asthma ABPA group only), blood routine test, Aspergillus-specific IgE and IgG detection, total immunoglobulin IgE, allergen detection, etc. Dust was collected indoors (bedrooms), outdoor (balconies) and on the surface of air conditioners or fans (if applicable) in the subject's living environment, and environmental data such as ambient temperature, humidity, and particulate matter concentration were recorded. 18S rRNA technology was used for sputum and dust fungus detection, and ELISA was used for asthmatitis symptomatic markers, which assess the impact of fungal infections on the disease. Follow-up for each subject 6 months, 6 months after enrollment, the patient's symptom changes, acute exacerbations/exacerbations, and prognosis were recorded, and relevant questionnaire scores were completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-80 years old (including 18 and 80 years old), gender and race are not limited;
2. No history of asthma, ABPA, or other chronic respiratory diseases.
3. No history of allergic diseases, such as allergic rhinitis, eczema, or food allergies.
4. Pulmonary function is normal or close to the normal range.
5. Laboratory testing:

1. Blood routine: High sensitivity C-reactive protein, white blood cells, neutrophils, lymphocytes, and monocytes are all within the normal range.

Allergen testing: IgE levels for common allergens such as dust mites, cat hair, dog hair, cockroaches, mold, and pollen are normal or close to the normal range.

Exclusion Criteria:

1. Suffering from bronchial asthma ABPA、 Bronchiectasis or other respiratory diseases: chronic obstructive pulmonary disease, active pulmonary tuberculosis, pulmonary embolism, lung cancer, pneumothorax, hemoptysis, pulmonary arterial hypertension, interstitial lung disease, etc;
2. Cancer patients who suffer from serious other systemic diseases, such as myocardial infarction, stroke, hypertensive crisis or refractory hypertension, severe arrhythmia, heart failure, aortic aneurysm, liver failure, renal failure, hematological disorders, etc., and have recently been discovered or are currently receiving treatment;
3. Four weeks prior to enrollment, systemic use of antibiotics, antifungal drugs, immunosuppressants, cytotoxic agents, hormones, etc;
4. Other individuals with contraindications for induced sputum testing:

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No bronchial asthma ABPA、 Healthy individuals aged 18-80 with bronchiectasis or other respiratory diseases
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory fungi | Baseline
  Analysis of sputum samples from patients with bronchial asthma, ABPA, and bronchiectasis using 18sRNA sequencing fungal diversity and abundance in liquid samples.

SECONDARY OUTCOMES:
Environmental fungi | Baseline
  Assess fungal diversity and abundance in the environment, including indoor (bedroom), outdoor (balcony), and air conditioning or fan surfaces (if applicable).
FEV1（Forced Expiratory Volume in 1 second） | Baseline
  Pulmonary function FEV1 index was evaluated in liters (L). It refers to the volume of air exhaled in the first second by the subject exhaling at the fastest rate after the maximum inspiration.
PEF （Peak Expiratory Flow） | Baseline
  PEF is measured in liters per minute (L/min). It refers to the maximum flow rate that can be achieved when exhaling at the fastest speed after the maximum inspiration. This indicator can reflect how open the airway is.
MMEF75/25（Maximal Mid-Expiratory Flow between 75% and 25% of FVC） | Baseline
  MMEF75/25 is measured in liters per minute (L/min). This is the average expiratory flow rate over the course of 75% to 25% of the forced expiratory volume. It is primarily used to assess the function of the small airways.
FVC （Forced Vital Capacity） | Baseline
  FVC is measured in liters (L). It is the maximum volume of air that can be exhaled by exhaling forcefully as fast as possible after the maximum inhalation. This indicator reflects the ventilatory function of the lungs. FVC is generally around 3.5 - 5 L in normal adult males and slightly lower in females. FVC can be used to assess the elasticity of the lungs, the patency of the airways, etc.
FEV1/FVC （Forced Expiratory Volume in 1 second to Forced Vital Capacity Ratio） | Baseline
  The unit of FEV1/FVC is %. It is mainly used to determine if there is an airflow obstruction. Normally, FEV1/FVC should be greater than 70%.
Number of Acute Exacerbations | Baseline, 6-month follow-up.
  The unit of Number of Acute Exacerbations is number of events. Total count of acute exacerbations experienced by participants.
Severity Grading of Acute Exacerbations | Baseline, 6-month follow-up.
  The unit of Severity Grading of Acute Exacerbations is units on a severity scale. Severity of each acute exacerbation categorized by a standardized scale (e.g.mild/moderate/severe or graded numerically, such as Grade 1-3).
Frequency of Emergency Department Visits | Baseline, 6-month follow-up.
  The number of emergency department visits due to acute exacerbations of Asthma, ABPA, and Bronchiectasis will be tracked using patients' self-reports and verified through medical records. This measure helps to evaluate the severity of the diseases.
Frequency of Hospitalizations | Baseline, 6-month follow-up.
  The number of people hospitalized due to acute exacerbations of Asthma, ABPA, and Bronchiectasis will be recorded, including detailed information such as the length of hospital stay and the treatments administered.
The use of emergency medication | Baseline, 6-month follow-up.
  Including the types of emergency drugs (such as salbutamol), as well as the dosage (number of presses), frequency of use, and duration of use
Occurrence of Respiratory Failure | Baseline,6-month follow-up.
  Documentation of respiratory failure events during hospital stays, including clinical criteria for diagnosis and management details.
Use of Non-Invasive Ventilation | Baseline,6-month follow-up.
  Documentation of the use of non-invasive ventilation during hospitalization, including indications and duration of use.
ICU Admission and Intubation | Baseline,6-month follow-up.
  Records of ICU admissions and whether intubation was required during hospitalization, including associated clinical details.
Systemic Steroid Use | Baseline,6-month follow-up.
  Documentation of systemic corticosteroid use during hospital stays, including dosage and duration.
Length of Hospital Stay | Baseline, 6-month follow-up.
  Total duration of each hospital stay will be recorded to assess the impact of the intervention on hospitalization length.
Asthma Control Questionnaire | Baseline, 6 month follow-up.
  In the asthma and ABPA research groups, the Asthma Control Questionnaire (ACQ) will be used to evaluate the control of asthma symptoms. ACQ is a validated questionnaire, with each question scoring 0-6 points. The average score will be calculated, with ≤ 0.75 indicating good control, 0.75-1.5 indicating partial control, and>1.5 indicating uncontrolled
AQLQ （Asthma Quality of Life Questionnaire） Score | Baseline, 6 month follow-up.
  The Asthma Quality of Life Questionnaire is used to evaluate the quality of life of asthma patients. The scoring range is 1 - 7 points. The higher the score, the better the quality of life.
FACED Score | Baseline, 6 month follow-up.
  FACED Score includes Forced Expiratory Volume in 1 second (FEV1)、Age、 Chronic colonization by Pseudomonas aeruginosa (PA)、Extension (number of pulmonary lobes affected)、Dyspnea (mMRC score).It is used to assess the severity of bronchiectasis. The scoring range is from 0 to 10 points. Grade classification: 0 - 2 points: Mild. 3 - 5 points: Moderate. 6 - 10 points: Severe.
Borg rating | Baseline, 6 month follow-up.
  The Borg score is used to evaluate the degree of respiratory distress in patients with bronchiectasis, measuring their perceived physical activity or intensity using numbers. Subjective fatigue and respiratory distress are quantified on a 0-10 point scale, with higher scores indicating more severe respiratory distress
BEST （Bronchiectasis Evaluation Score for Treatment)）Score | Baseline, 6 month follow-up.
  The BEST Score is used to assess the symptoms of dyspnea and cough. The scoring range is from 0 to 10 points. Grade classification: 0 - 2 points: Mild. 3 - 5 points: Moderate. 6 - 10 points: Severe.
CAT（COPD Assessment Test） Score | Baseline, 6 month follow-up.
  A tool used in the bronchiectasis group to assist in assessing the severity and quality of life of patients with bronchiectasis. The rating range is 0-10 points. Grade classification: 0-2 points: Mild; 3-5 points: moderate; 6-10 points: severe.
Electronic X Asthma Control Test | Baseline, 6 month follow-up.
  In the bronchiectasis group, it is used to assist in evaluating the daily condition of bronchiectasis patients, such as symptoms, sputum volume, and nighttime awakening. The score ranges from 0 to 100, with higher scores indicating poorer disease control.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang Recruiting, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No